CLINICAL TRIAL: NCT01940263
Title: Effects of Purified Anthocyanin on Oxidative and Inflammatory Markers in Subjects With Nonalcoholic Fatty Liver Disease: A Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Purified Anthocyanin and Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shaoguan University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SGU-02; 81372994 (Other: National Natural Science Foundation of China)
Record Dates: First submitted 2013-09-02; First posted 2013-09-12 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: oxidative stress; dyslipidemia; inflammation; apoptosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Dyslipidemias; Inflammation | interventions — Anthocyanins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo 320 mg daily for twelve weeks
  Interventions: Dietary Supplement: Placebo
- Anthocyanin (Experimental): Drug: MEDOX (natural purified anthocyanin) anthocyanin 320 mg daily for twelve weeks.
  Interventions: Dietary Supplement: Anthocyanin

INTERVENTIONS:
Dietary Supplement: Anthocyanin
  Other Names: MEDOX (natural purified anthocyanin); http://www.medox.no/english
  Arms: Anthocyanin
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Oxidative stress and inflammation are involved in the pathogenesis of non-alcoholic fatty liver disease (NAFLD). Anthocyanins from different plant foods have been shown to improve features of experimental NASH, such as oxidative stress, dyslipidemia, liver steatosis, and inflammation in rodents. The purpose of this study is to investigate whether purified anthocyanin supplementation beneficially alters oxidative, inflammatory, and apoptotic biomarkers in adults with features of NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* BMI [body weight divided by height squared (in kg/m2)] > 23,
* lack of excessive alcohol ingestion confirmed by careful questioning by the primary physician and dietitians (consumption of less than 70 g alcohol in female and 140 g in male per week), and
* the presence of two of the three following diagnostic criteria of the fatty liver disease: increased hepatic echogenicity compared to the spleen or the kidneys, blurring of liver vasculature and deep attenuation of the ultrasonographic signal.

Exclusion Criteria:

* overuse of alcohol,
* viral hepatitis,
* type 1 or 2 diabetes,
* gastrointestinal or connective diseases,
* chronic pancreatitis,
* liver cirrhosis,
* kidney stones, or renal failure;
* use of acetyl-salicylic acid or other antiplatelet drugs, statins of fibrates, oral hypoglycemic drugs, nitrates, nonsteroidal antiinflammatory drugs, corticosteroids, or drugs interfering with coagulation;
* supplementation with vitamins or antioxidants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Biomarkers related to oxidative stress | Twelve weeks
  plasma total antioxidant capacity; plasma levels of protein carbonyl groups

SECONDARY OUTCOMES:
Biomarkers related to inflammation | Twelve weeks
  tumor necrosis factor alpha; interleukin-8; high sensitive C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Wenhua Ling, Ph.D, Study Director — Sun Yat-sen University
Locations (1):
- Shaoguan University, Shaoguan, Guangdong, China

REFERENCES:
- [Derived] Zhang PW, Chen FX, Li D, Ling WH, Guo HH. A CONSORT-compliant, randomized, double-blind, placebo-controlled pilot trial of purified anthocyanin in patients with nonalcoholic fatty liver disease. Medicine (Baltimore). 2015 May;94(20):e758. doi: 10.1097/MD.0000000000000758. PMID 25997043
- [Derived] Liu Y, Chen H, Wang J, Zhou W, Sun R, Xia M. Association of serum retinoic acid with hepatic steatosis and liver injury in nonalcoholic fatty liver disease. Am J Clin Nutr. 2015 Jul;102(1):130-7. doi: 10.3945/ajcn.114.105155. Epub 2015 May 6. PMID 25948673